CLINICAL TRIAL: NCT01176851
Title: Pharmacokinetic, Randomized, Open-label, Single-dose, 3-way Cross-over Study of Intravenous and Inhaled Glycopyrrolate With or Without Charcoal Block Ingestion in Healthy Volunteers.
Brief Title: Biopharmaceutical Study of Glyco pMDI With or Without Charcoal Block vs IV Bolus in Healthy Volunteers
Acronym: Gly1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Martine Cartier, Head of Clinical Operations, Chiesi Farmaceutici SpA
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CCD-0915-PR-0031
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Healthy
Keywords: None (study in healthy volunteers)
MeSH Terms: interventions — Glycopyrrolate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Glyco pMDI (Experimental): Glyco pMDI 100 µg
  Interventions: Drug: Glycopyrrolate
- Glyco pMDI Charcoal (Experimental): Glyco pMDI 100 µg + charcoal block
  Interventions: Drug: Glycopyrrolate
- Glyco IV injection (Active Comparator): Glyco solution for injection 100 µg
  Interventions: Drug: Glycopyrrolate

INTERVENTIONS:
Drug: Glycopyrrolate — Single administration of Glyco pMDI 100 µg
  Other Names: CHF 5259
  Arms: Glyco pMDI
Drug: Glycopyrrolate — Single administration of Glyco pMDI 100 µg after charcoal ingestion
  Other Names: CHF 5259
  Arms: Glyco pMDI Charcoal
Drug: Glycopyrrolate — Single intravenous injection of glycopyrrolate 100 µg
  Other Names: Robinul Injection
  Arms: Glyco IV injection

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics, the absolute bioavailability and the lung bioavailability of inhaled Glyco pMDI.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females healthy volunteers aged 18-65 years;
2. Written informed consent obtained before the first trial related activity.
3. Able to understand the study procedures, the risks involved and ability to be trained to use the devices correctly.
4. Body Mass Index (BMI) between 18.0 and 32.0 kg/m2;
5. Non- or ex-smokers who smoked < 5 pack years;
6. Good physical and mental status;
7. Normal blood pressure and heart rate;
8. Electrocardiogram (ECG)considered as normal;
9. Results of laboratory tests within the normal ranges.
10. Lung function measurements within the normal ranges.

Exclusion Criteria:

1. Blood donation (equal or more than 450 ml) or blood loss less than 8 weeks before inhalation of the study medication;
2. Pregnant or lactating women or women of childbearing potential, UNLESS they are using one or more of the acceptable methods of contraception. Male subjects not willing to use an acceptable method of contraception.
3. Positive HIV1 or HIV2 serology;
4. Positive results from the Hepatitis serology which indicates acute or chronic Hepatitis B or Hepatitis C;
5. Unsuitable veins for repeated venipuncture;
6. History of substance abuse or drug abuse within 12 months prior to screening visit or with a positive urine drug screen at screening;
7. Clinically relevant abnormal laboratory values suggesting an unknown disease and requiring further clinical investigation;
8. Clinically significant and uncontrolled cardiac, hepatic, renal, gastrointestinal, endocrine, metabolic, neurologic, or psychiatric disorder that may interfere with successful completion of this protocol;
9. Participation in another clinical trial less than 8 weeks prior to inhalation of the study medication; participation in another clinical trial using radioactive material within 1 calendar year;
10. History of hypersensitivity to M3 Antagonists or any of the excipients contained in any of the formulations used in the trial;
11. Any drug treatment, including prescribed or OTC medicines as well as vitamins, homeopathic remedies etc, taken in the 14 days (2 months for enzyme-inducing or enzyme-inhibiting drugs e.g., glucocorticoids, phenobarbital, isoniazid) preceding the first intake of the study drug, with the exception of occasional paracetamol (maximum 2 g per day with a maximum of 10 g per 14 days for mild non-excluding conditions).
12. Treatment within the previous 3 months with any drug known to have a well defined potential for hepatotoxicity (e.g. isoniazide, nimesulide, ketoconazole).
13. Subjects who refuse to abstain from alcohol or caffeine containing foods or beverages or grapefruit containing foods or beverages from 48 hour prior to the first intake of study medication and for the entire duration of the study.
14. Heavy caffeine drinker.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Plasma and urine pharmacokinetics of glycopyrrolate | over 24 h post dose

SECONDARY OUTCOMES:
Lung function parameters | over 24 h post dose
Cardiovascular parameters | over 24 h post dose
Clinical chemistry and haematology, urinalysis | over 24 h post dose
Adverse Events | during the whole study period

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, MD, Principal Investigator — Medicines Evaluation Unit
Locations (1):
- Medicines Evaluation Unit, Manchester, United Kingdom

REFERENCES:
- See also: CSR Synopsis available in the Chiesi Clinical Study Register — https://www.chiesi.com/clinic/CSR_Synopsis_CCD-0915-PR-0031.pdf